CLINICAL TRIAL: NCT04752891
Title: Assessment of an App Based on Artificial Intelligence for Purulent Acute Otitis Media (AOM) Diagnosis in a a Pediatric Emergency Department
Brief Title: Assessment of an App Based on Artificial Intelligence for Purulent AOM Diagnosis in a Pediatric Department
Acronym: OMA-IA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-HPNCL-07
Record Dates: First submitted 2021-02-02; First posted 2021-02-12 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Otitis Media, Suppurative
MeSH Terms: conditions — Otitis Media, Suppurative | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AOM diagnosis with app (Experimental)
  Interventions: Other: AOM diagnosis with app
- AOM diagnosis without app (Other)
  Interventions: Other: AOM diagnosis without app

INTERVENTIONS:
Other: AOM diagnosis with app — the diagnosis made by a senior physician using a traditional otoscope. the diagnosis made by the junior physician using an otoendoscope fixed on a connected smartphone
  Arms: AOM diagnosis with app
Other: AOM diagnosis without app — the diagnosis made by a senior physician and by the junior physician, using a traditional otoscope
  Arms: AOM diagnosis without app

SUMMARY:
Otitis media (OM) is one of the most common childhood infections and is a major cause of morbidity in children and results as being the first cause of antibiotic prescription among children in developed countries . An artificial intelligence-based tool could help physicians refine their diagnosis

DETAILED DESCRIPTION:
Ear infections in children are very common, particularly acute otitis media (AOM) which represents the first reason for visiting physicians and for antibiotic prescription in children in developed countries. However, the diagnosis is not easy because of the narrowness of the ear canal, the discomfort of the child during the otoscopic exam. Moreover, the accuracy of the AOM diagnosis depends on the subjectivity of the physician mostly. This can result in an misdiagnosis and inappropriate treatment with, as a result, the emergence of multi-resistant germ.

Artificial intelligence (AI) in medicine is booming and has already proven its worth in terms of prevention, monitoring and diagnosis. I-Nside, an app based on Artificial Intelligence is able to make automatic diagnosis of many ear pathologies, after capturing picture of any eardrum using an otoendoscope fixed on a connected smartphone (SmartScope®).

Therefore, the investigators aim to assess the accuracy of AOM diagnosis the existing app, by comparing the inter-rater agreement between the diagnosis made by a senior physician using a traditional otoscope (considered as "gold standard" ) and the one made by a junior physician using the app

ELIGIBILITY:
Inclusion Criteria:

Child under 18 years Presenting signs that may suggest acute otitis media (fever, earache, purulent otorrhea) For which the informed written consent of, at least, one of the two parents or the holder of parental authority has been obtained

Exclusion Criteria:

A sign (s) of vital distress Trans-tympanic drains

-

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 203 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
diagnosis of purulent Acute Otitis Media (AOM) made by junior physicians using the i-Nside application associated with Smartscope® | at inclusion
  diagnosis of purulent AOM is made on an inflammatory aspect of the eardrum with retrotympanic effusion, exteriorized (otorrhea) or not (opacity, effacement of reliefs or bulging, disappearance of the light triangle).
diagnosis of purulent Acute Otitis Media (AOM) made by senior physicians using a standard otoscope | at inclusion
  diagnosis of purulent AOM is made on an inflammatory aspect of the eardrum with retrotympanic effusion, exteriorized (otorrhea) or not (opacity, effacement of reliefs or bulging, disappearance of the light triangle)

SECONDARY OUTCOMES:
rate of misdiagnoses of purulent Acute Otitis Media (AOM) with and without the use of the application | at inclusion
  a misdiagnosis is measured by a discordant diagnosis of the juniors compared to the seniors considered as the Gold Standard for the AOM diagnosis
collection risk factors for a discrepancy in the diagnosis of purulent AOM | at inclusion
  collection data of age of patients,pain requiring analgesia, period of the day of diagnosis (morning, afternoon,night)
satisfaction of junior physicians regarding the use of the app | through study completion, an average of 1 year
  a questionnaire will be given at the end of the study. The questions relate to the use of the application and its perceived usefulness by practitioners. Satisfaction will be assessed by a Lickert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Pédiatrique de Nice CHU Lenval, Nice, France